CLINICAL TRIAL: NCT06499155
Title: Comparison of the Clinical Efficacy of Cyanoacrylate Tissue Adhesive With Suture in the Treatment of Gingival Recession
Brief Title: Comparison of Cyanoacrylate Tissue Adhesive With Suture in the Treatment of Gingival Recession
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Kevser Yildirim, Research Assistant, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: periacrylinCTG
Record Dates: First submitted 2024-03-28; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Gingival Recession
Keywords: connective tissue graft; coronally advanced flap; periacryl
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- tissue adhesive group (Active Comparator): Only tissue adhesive will be used for primary closure of the donor area. After the flap is closed with sutures in the recipient area, it will be supported with tissue adhesive.
  Interventions: Device: Use of periacryl in gingival recession closure procedures; Procedure: Use of sutures in gingival recession closure procedures
- suture group (Active Comparator): The donor and recipient areas will be closed with sutures.
  Interventions: Device: Use of periacryl in gingival recession closure procedures; Procedure: Use of sutures in gingival recession closure procedures

INTERVENTIONS:
Device: Use of periacryl in gingival recession closure procedures — Unlike the traditional procedure, periacryl tissue adhesive will be used in both the recipient and donor areas.
Procedure: Use of sutures in gingival recession closure procedures — Both recipient and donor areas will be closed with traditional suturing techniques.

SUMMARY:
The aim of this randomized controlled clinical study was to determine the effects of gingival recession closure procedures performed with tissue adhesive and suture on gingival thickness, To evaluate the effect on the amount of gingival recession, keratinized tissue amount, clinical attachment level, probing pocket depth, papilla width and height, root coverage rate, wound healing, visual analogue scale, gingival index and plaque index.

The main questions it aims to answer are:

* Does the use of tissue adhesive in gingival recession closure procedures affect tissue healing in the recipient area?
* Does the use of tissue adhesive in gingival recession closure procedures affect tissue healing in the donor area? Participants will be informed about the study and the procedures to be performed, and the patients will continue their routine follow-up.

DETAILED DESCRIPTION:
Gingival recession is known as the apical displacement of the gum from the cement-enamel junction. Various root coverage procedures have been successfully performed to prevent recession, correct aesthetic problems, help control plaque, and reduce dentin hypersensitivity.

The ultimate goal of the root coverage procedure is to prevent, correct or eliminate the recession defect with an appearance compatible with the adjacent soft tissues following healing and with minimal probing depth.

The aim of this study is to evaluate the clinical effectiveness of fixing the donor area with periacryl tissue adhesive instead of suture and supporting the sutures placed on the flap in the recipient area with periacryl tissue adhesive in modified coronally placed flap operations performed in combination with subepithelial connective tissue graft in patients with Miller class I and II gingival recession. to evaluate and compare with the classical technique using only sutures.

This study is planned to be conducted on 40 individuals aged between 18-65. Patients who do not have any systemic disease, do not smoke or drink alcohol, are not pregnant or breastfeeding, have not used antibiotics in the last 6 months, and do not use regular medication will be included in the study.

In this study, patients will be divided into 2 groups according to whether they use periacryl or not.

This study is planned prospectively and the initial, 1st, 3rd, 6th and 12th month follow-up measurements of the patients who will be treated in our clinic will be evaluated. In the measurements, gingival recession parameters including probing depth, clinical attachment level and recession depth, keratinized tissue width and gingival thickness will be evaluated. In multiple gingival recessions, plaque index and gingival index will be obtained from three points: mesial, distal and midpoints; The plaque index will be calculated according to the criteria determined by Silness and Loe, while the gingival index will be calculated according to the criteria determined by Loe and Silness.

On postoperative days 1, 3, and 7, patients will be asked to fill out a table in which they can score their subjective complaints of pain, burning sensation, and discomfort in the surgical area on a personal pain scale (VAS) ranging from 0 (not at all) to 100 (very severe).

In this study, the physician; When removing stitches 2 weeks after surgery, the wound healing index will be filled in for each tooth individually, evaluated according to Huang's criteria:

In this randomized controlled clinical study, it was determined in which of 40 patients periacryl tissue adhesive would be used and in which suture; It will be determined by computer-assisted randomization method (www.randomizer.org). All surgical procedures and measurements will be performed by the same clinician.

The primary endpoint was 6-month clinical follow-up of gingival recession closure procedures; The aim is to determine the effect on wound healing and tissue thickness in the donor area and on the root surface coverage rate and tissue thickness in the recipient area.

surgical procedure Root surfaces in gingival recession areas will be smoothed using Gracey curettes.

Submarginal incisions will be made in the interdental areas and intrasulcular incisions will be made around the teeth with recession defects. Half-full-half thickness flap incisions will be applied in the corona-apical direction.

No vertical relaxing incision will be made, and the papilla adjacent to the relevant tooth will be de-epithelialised to create a connective tissue bed. In surgical areas, the previously prepared subepithelial connective tissue graft will be fixed to the periosteum using 5-0 resorbable suture. The flap will be designed to be relieved by an incision of the periosteum and positioned coronally without tension. The area will be closed with 5-0 non-resorbable stitches and hemostasis will be achieved by applying light finger pressure for 4 minutes. Sutures will be supported with periacryl tissue adhesive in half of the patients.

The palatal donor area will be measured with a periodontal probe to ensure that the soft tissue thickness is at least 3 mm, and a parallel incision will be made in the donor area, usually in the palatal area between the maxillary first molar and the maxillary canine, staying at least 2 mm away from the tooth edge. A vertical relaxing incision will be applied to remove the subepithelial connective tissue graft from the palate. The palate will be sutured with 4-0 absorbable suture or secured with periacryl tissue adhesive. Before the connective tissue is placed in the recipient area, the fatty and secretory tissue and the band-shaped epithelium overlying the connective tissue will be removed using scissors.

Stitches will be removed 14 days after surgery. Interdental care will begin approximately 2 weeks after the stitches are removed, patients will be asked to come for routine control visits 1, 3, 6 months after the surgery, and clinical measurements and/or photographs will be taken during the control visits.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers between the ages of 18-65
* Absence of any systemic disease such as endocrine disease, nephrotic syndrome, chronic renal disease and cardiovascular disease
* Not having uncontrolled diabetes mellitus with HbA1c>7,
* Not smoking and not having any blood diseases,
* Not having used antibiotics in the last 6 months for any reason,
* There must be no previous surgical procedure in the selected areas.
* The presence of periodontal pockets not exceeding 3 mm in size on the treated teeth; No occlusal trauma to teeth
* Having at least 20 teeth in the mouth
* People who are not pregnant or breastfeeding and who are not taking any regulatory medication.
* Patients who applied to the periodontology clinic with various periodontal problems and received an indication for connective tissue graft operation due to receding gums
* There is no systemic condition that may prevent surgical application.
* Not using drugs systemically

Exclusion Criteria:

* Not to be in inclusion criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the effect of periacryl on wound healing in the donor area with a visual analog scale | 6 months
  In clinical follow-ups of gingival recession closure procedures; Wound healing in the donor area will be monitored with the help of a visual analog scale filled in by the patient.
Determining the effect of periacryl on the root surface closure rate in the recipient area by proportioning the amount of root closure to the initial recession amount. | 6 months
  In clinical follow-ups of gingival recession closure procedures; Root surface closure rate in the recipient area; After the procedure, the amount of closure obtained in millimeters is divided by the initial amount of gingival recession to obtain a percentage value. Using these data, the effect of periacryl on the root surface closure rate will be determined.
The effect of periacryl on the tissue thickness obtained after the procedure in the recipient area | 6 months
  In clinical follow-ups of gingival recession closure procedures; The increase in keratinized tissue thickness obtained in the recipient area will be measured in millimeters using the who probe. The data obtained will be compared to the initial keratinized tissue thickness amounts. In this way, the effect of periacryl on the increase in keratinized tissue in the recipient area will be observed.

CONTACTS AND LOCATIONS:
Overall Officials: KEVSER YILDIRIM, RA, Principal Investigator — Necmettin Erbakan University